CLINICAL TRIAL: NCT01084499
Title: Bioequivalence Study of YUHAN Letrozole 2.5 mg Tablets
Brief Title: Bioequivalence Study of Letrozole 2.5 mg Tablets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: YCD143
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Results first posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Healthy
Keywords: Healthy Subjects
MeSH Terms: interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Femara First, Then Peratra (Sequence 1) (Experimental): Participants first receives a branded letrozole (reference - Femara), then a generic letrozole (test - Peratra). Each treatment period is separated by a 5-week washout period.
  Interventions: Drug: Femara (Sequence 1); Drug: Peratra (Sequence 1)
- Peratra First, Then Femara (Sequence 2) (Experimental): Participants first receives a generic letrozole (test - Peratra) , then a branded letrozole (reference - Femara). Each treatment period is separated by a 5-week washout period.
  Interventions: Drug: Femara (Sequence 2); Drug: Peratra (Sequence 2)

INTERVENTIONS:
Drug: Femara (Sequence 1) — Participant who is assigned to the Sequence 1 first receive Femara, then a Peratra. Each treatment period is separated by a 5-week washout period.
  Other Names: Femara Tab.[Letrozole 2.5mg]
  Arms: Femara First, Then Peratra (Sequence 1)
Drug: Peratra (Sequence 1) — Participant who is assigned to the Sequence 1 first receive Femara, then a Peratra. Each treatment period is separated by a 5-week washout period.
  Other Names: Peratra Tab.[Letrozole 2.5mg]
  Arms: Femara First, Then Peratra (Sequence 1)
Drug: Femara (Sequence 2) — Participant who is assigned to the Sequence 2 first receive Peratra, then a Femara. Each treatment period is separated by a 5-week washout period.
  Other Names: Femara Tab.[Letrozole 2.5mg]
  Arms: Peratra First, Then Femara (Sequence 2)
Drug: Peratra (Sequence 2) — Participant who is assigned to the Sequence 2 first receive Peratra, then a Femara. Each treatment period is separated by a 5-week washout period.
  Other Names: Peratra Tab.[Letrozole 2.5mg]
  Arms: Peratra First, Then Femara (Sequence 2)

SUMMARY:
Bioequivalence

DETAILED DESCRIPTION:
The purpose of this study was to determine the bioequivalence of letrozole 2.5 mg tablets after administration of single doses to normal healthy Korean subjects under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers in the age between 19 to 55 years old
* Subjects were neither congenital nor chronic diseases.
* Subjects were selected after passing a clinical screening procedure that included a physical examination and laboratory tests.
* Availability of subject for the entire study period and willingness to adhere to protocol requirements, as evidenced by a signed Informed Consent Form.

Exclusion Criteria:

* Any history of a clinical condition which might affect drug absorption, distribution, metabolism or excretion or might be risk factors, e.g. clinically significant disorder in heart, liver, respiratory system, liver, kidney, gastrointestinal system and CNS
* Had a history of myocardial infarction, stroke, hypertension, arrhythmia, coronary artery disease, disease of neuropsychiatry, gastrointestinal system surgery (excluding appendectomy, herniotomy)
* Current clinically significant disorder in history taking or physical examination
* Acute disease within 14 days preceding the first application of study medication
* Had an relevant allergic disease
* Had history of hypersensitivity to drugs or any food
* Positive for Hepatitis B antigen, Hepatitis C antibody, HIV antibody, or High Quality Syphilis Reagin Test
* Excessive caffeine, alcohol intake and smoker(caffeine>5 units/day, alcohol>3 units/day(1 unit = pure alcohol 10ml), cigarettes> 20 cigarettes /day)
* Subjects who excessive alcohol intake or drug which affect drug metabolism enzyme intake within 30 days preceding study
* History of drug abuse or positive for urinary testing of drugs abuse (amphetamine, barbiturates, cocaine, opioids, benzodiazepines etc.)
* Has donated whole blood within 60days or apheresis within 14days preceding the first application of study medication
* Received other investigational drug within 60days preceding the first application of study medication
* Taken any herbal medicine within 30days, prescription medication within 14 days or over-the-counter drug (except for vitamins, minerals) within 10days preceding the first application of study medication (might affect this study or safety of subjects as judged by the investigator)
* Subjects couldn't eat ASAN MEDICAL CENTER standard meal or were unsuitable for this study as judged by investigators

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyeong-seok Lim, MD, PhD, Principal Investigator — Asan Medical Center

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study period: Jan 2009 ~ May 2009
Groups:
- Femara First, Then Peratra (Sequence 1): Participants first received a branded letrozole (reference - Femara), then a generic letrozole (test - Peratra). Each treatment period was separated by a 5-week washout period.
- Peratra First, Then Femara (Sequence 2): Participants first received a generic letrozole (test - Peratra), then branded letrozole (reference - Femara). Each treatment period was separated by a 5-week washout period.
Period: Overall Study
Arm/Group | Femara First, Then Peratra (Sequence 1) | Peratra First, Then Femara (Sequence 2)
Started | 13 (First Intervention (Sequence 1) : Femara (1 Day)) | 13 (First Intervention (Sequence 2) : Peratra (1 Day))
Washout (5 Weeks) | 13 | 13
Completed | 13 (Second Intervention (Sequence 1) : Peratra (1 Day)) | 13 (Second Intervention (Sequence 2) : Femara (1 Day))
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Peratra First, Then Femara (Sequence 2): Participants first received a generic letrozole (test - Peratra), then a branded letrozole (reference - Femara). Each treatment period was separated by a 5-week washout period.
- Total: Total of all reporting groups
Arm/Group | Femara First, Then Peratra (Sequence 1) | Peratra First, Then Femara (Sequence 2) | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 28.8 (4.8) | 27.5 (4.1) | 28.1 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Letrozole : AUC0-tz
Description: Area Under the Concentration-time Curve of Letrozole in Plasma Over the Time Interval From 0 to the Time of the Last Quantifiable Data Point.
Time Frame: Predose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 48, 96, 168, 312 hrs after drug administration
Measure: Mean (Standard Deviation); unit: ng•hr/mL
Groups:
- Peratra: The group of participants who were administered Peratra.
- Femara: The group of participants who were administered Femara.
Arm/Group | Peratra | Femara
Number analyzed (Participants) | 26 | 26
ng•hr/mL | 2074.71 (826.15) | 2094.63 (870.79)

2. Primary Outcome: Letrozole : Cmax
Description: Maximum Measured Concentration of Letrozole in Plasma
Time Frame: Predose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 48, 96, 168, 312 hrs after drug administration
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Peratra | Femara
Number analyzed (Participants) | 26 | 26
ng/mL | 35.38 (6.66) | 38.13 (7.03)

ADVERSE EVENTS:
Time Frame: 10 Weeks (1) First Intervention : 2 Weeks (Blood samples were obtained before dosing and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 48, 96, 168, and 312 hours after oral administration of 2.5 mg of letrozole) (2) Washout : 5 Weeks (3) Second Intervention : 2 Weeks (4) Last safety profile assessment : 1 Weeks
Arm/Group | Peratra | Femara
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 8/26 | 4/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Peratra (N=26) | Femara (N=26)
Abdominal Discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Asthenia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1/13 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Ankle sprain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Blood Bilirubin Increased (Investigations) | 1 (1) | 1 (1)
Blood Triglyceride Increased (Investigations) | 1 (1) | 1 (1)
Creatine Kinase Increased (Investigations) | 1 (1) | 1 (1)
Blood Lactate Dehydrogenase Increased (Investigations) | 1 (1) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0)
Blood Calcium Increased (Investigations) | 1 (1) | 0 (0)
Urinary Occult Blood Positive (Investigations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study shall be owned by the Sponsor. The results of this study can be published in journals with the consent of the Sponsor, and the Sponsor can also request the presentation of the results to the investigator(s).